CLINICAL TRIAL: NCT01047189
Title: Adherence to ZIANA (Clindamycin Phosphate 1.2% With Tretinoin 0.025%)Gel Compared to Generic Topical Clindamycin Plus Generic Topical Tretinoin in Subjects With Mild to Moderate Acne Vulgaris
Brief Title: Adherence to Study Medication Compared to Generic Topical Clindamycin Plus Generic Topical Tretinoin in Subjects With Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00007137
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Acne Vulgaris
Keywords: Mild to moderate acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; clindamycin, tretinoin drug combination; Clindamycin; Gels; Tretinoin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Ziana gel (clindamycin phosphate 1.2% and tretinoin 0.025%) applied once daily for 12 weeks
  Interventions: Drug: clindamycin phosphate 1.2% and tretinoin 0.025%
- 2 (Active Comparator): Generic clindamycin 1% gel plus tretinoin 0.025% cream
  Interventions: Drug: clindamycin 1% gel; Drug: tretinoin 0.025% cream

INTERVENTIONS:
Drug: clindamycin phosphate 1.2% and tretinoin 0.025% — applied once daily for 12 weeks
  Other Names: Ziana
  Arms: 1
Drug: clindamycin 1% gel — Topical clindamycin applied each morning for 12 weeks
  Arms: 2
Drug: tretinoin 0.025% cream — Tretinoin 0.025% cream each evening for 12 weeks
  Arms: 2

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of two different types of topical acne medication. This study will help to determine if one combined medication results in better acne improvement than two separate medications for acne.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females 12 years of age or older with a diagnosis of mild to moderate acne vulgaris.
* Subjects must sign written informed consent and agree to come for all study visits.

Exclusion Criteria:

* Use of experimental drugs within 1 month prior to initiation of study therapy.
* Pregnant and nursing females will not be allowed in the study, and females of childbearing potential will have a pregnancy test at baseline. Females of childbearing potential must agree to use approved birth control methods for the duration of the study.
* Use of systemic retinoids within 2 months of enrollment, use of any topical retinoids, systemic antibiotics, nicotinamide, systemic steroids or any other medication that may confound the results of the study within 1 month prior to start of the study
* Use of any other topical medications for acne, including cosmetics containing retinol, within 2 weeks prior to study entry.
* Any skin condition or disease that may require concurrent therapy or may confound the evaluation;
* History of hypersensitivity to any of the formulation components;
* Facial skin cancer or facial actinic keratosis;
* Use of any photosensitizing agents.
* Use of isotretinoin within the last 6 months.
* Chemical peels, microdermabrasion or laser resurfacing within 3 months of study entry.
* Crohns disease, ulcerative colitis, or have developed colitis with past antibiotic use.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Dermatology, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from IRB approved advertising and the Wake Forest University Health Sciences Dermatology Clinic
Groups:
- Ziana Gel: Ziana gel (clindamycin phosphate 1.2% and tretinoin 0.025%) applied once daily for 12 weeks
- Clindamycin Plus Tretinoin Applied Separately: Generic clindamycin 1% gel plus tretinoin 0.025% cream
Period: Overall Study
Arm/Group | Ziana Gel | Clindamycin Plus Tretinoin Applied Separately
Started | 13 | 13
Completed | 9 | 13
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziana Gel | Clindamycin Plus Tretinoin Applied Separately | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 2 | 9
  Between 18 and 65 years | 6 | 11 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 20.1 [13 to 35] | 26.2 [15 to 40] | 23.1 [13 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Measured Adherence to ZIANA Gel or Generic Topical Clindamycin 1% Gel Each Morning Plus Generic Topical Tretinoin 0.025% Cream Each Evening in Subjects With Mild to Moderate Acne
Description: Percentage of prescribed doses taken as measured by a Medication Event Monitoring System (MEMS) cap
Time Frame: 12 weeks
Population: All patients were analyzed up to end of treatment or last visit.
Measure: Median (Full Range); unit: Percent of doses
Arm/Group | Ziana Gel | Clindamycin Plus Tretinoin Applied Separately
Number analyzed (Participants) | 13 | 13
Percent of doses | 88 [13 to 115] | 61 [8 to 95]

2. Secondary Outcome: The Change (Dynamic Assessment) From Baseline to Week 12 (or End of Treatment) in Total Acne Lesion Count
Time Frame: Baseline to 12 weeks
Population: All patients were analyzed up to end of treatment or last visit.
Measure: Mean (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Ziana Gel | Clindamycin Plus Tretinoin Applied Separately
Number analyzed (Participants) | 13 | 13
percentage of lesions | -51 [-80 to -23] | -32 [-66 to 2]
Statistical Analysis 1: Comparison: Ziana Gel vs Clindamycin Plus Tretinoin Applied Separately; Test type: Superiority or Other; p = 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | Ziana Gel | Clindamycin Plus Tretinoin Applied Separately
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziana Gel (N=13) | Clindamycin Plus Tretinoin Applied Separately (N=13)
Burning sensation on facial skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No